CLINICAL TRIAL: NCT06822816
Title: Creation of a Video/Image Library of Annotated Full-length Endoscopy Procedures for the Development of Artificial Intelligence-empowered Endoscopy Quality Reporting and Educational Modules
Brief Title: Video/Image Library of Endoscopy Procedures for the Development of AI-empowered Endoscopy Quality Reporting and Educational Modules
Acronym: Videotheque
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Daniel Von Renteln, Gastroenterologist, Principal Scientist, MD, PhD, Centre hospitalier de l'Université de Montréal (CHUM)
Other Study IDs: 2023-10355/22.013
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Polyp of Colon; Artificial Intelligence (AI)
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to establish a video/image library dataset of complete endoscopy or partial colonoscopy procedures for patients with rectal cancer or inflammatory bowel disease (IBD). With this video/image library, the aims are:

* to develop and validate novel AI-empowered solutions to automatically detect and report endoscopy quality metrics
* to develop automated endoscopy reporting solutions, auditing, and educational tools for residents and fellows to enhance their endoscopy skills.

The hypothesis is that a heterogeneous video/image library will provide:

* comprehensive and robust source material to develop AI models
* real-time quality feedback at the end of an endoscopy procedure.

DETAILED DESCRIPTION:
The video/image library will be constructed by prospectively recruiting patients referred for endoscopy procedures for the upper or lower gastrointestinal tract diseases. Patients who have had a screening, surveillance, or diagnostic upper or lower endoscopy recorded as part of a research project at the CHUM will all be invited to participate in this banking.

A qualified and adequately trained study team representative will invite potential study patients to participate during and outpatient clinic visit, or at their arrival in the endoscopy unit on the day of the endoscopy.

Board-certified gastroenterologists, or trainees under supervison, will perform all upper or lower endoscopies at the CHUM. Patients will be prepared for endoscopies according to the most recent guidelines and current standards of care.

The complete or partial endoscopy will be video recorded and the data files will be saved without loss of image quality using Medicapture USB 300 (or equivalent) devices and stored locally in an on-site storage cloud. All videos will be recorded with timestamps burned into the recording. A research assistant will document all relevant informations and annotations during the procedure.

All esophagogastroduodenoscopies (EGDs) will be performed using the high-definition endoscopes. All findings (e.g., lesions, polyps, inflammations), diagnostics, and therapeutic procedures will be documented during EGDs.

The colonoscopies will be performed using high-definition colonoscopes equipped with image-enhanced techniques, or CAD systems, to provide real-time support to endoscopists to detect polyps of all sizes. If required, the endoscopists will be instructed to use white-light and narrow-band imaging to perform optical diagnosis (OD) for all 1-10mm polyps. An OD will first be performed without CADx, then CADx will be used to make a CAD-based OD.

After detecting a polyp and performing ODs, the endoscopists will remove all polyps using standard techniques. Endoscopists will annotate the withdrawal time before initiating a resection, and again when the resection is complete. All biopsy specimens and main polyp specimens will be sent to the institutional pathology laboratories (in separate jars) for histopathology assessments.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 y.o.
* indication of undergoing a screening, surveillance, diagnostic, or therapeutic upper (EGD) or lower (colonoscopy) endoscopy

Exclusion Criteria:

* Coagulopathy defined as an elevated INR ≥ 2.5
* Platelet count ≤ 50,000/mm3
* Emergency endoscopy
* Poor general health defined as the American Society of Anesthesiologists physical status class >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients presenting at the CHUM for an upper or lower endoscopy will be approached for this study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
EGD documented data | From enrollment to 14 days post-procedure
  For EGD procedures, the following data will be documented: the exact time to reach the GE junction, the diaphragmatic hiatus, body/fondus/antrum of stomach, duodenum, procedural time during EGD, complications (immediate and late: first 24h post-procedure and 14 days post-procedure, respectively), the use of a distal attachment cap, insufflation and desufflation, cardiac retroflexion for facilitating visualization of mucosa during EGD, the use of existing AI platforms that increase lesion detection (CADe) and classification (CADx), the AI classification (autonomous CADx diagnosis), the endoscopists' ODs without CADx, the endoscopists' ODs after seeing the diagnosis from CADx (CADx-assisted diagnosis), the performance of endoscopists (measured with detection rates such as ADR, AADR, SSLDR, PDR, or with detection counts such as APC).
Colonoscopy documented data | From enrollment to 14 days post-procedure
  For colonoscopy procedures, the following data will be documented: the exact time to reach the caecum, caecum intubation, the exact time of the visualisation of each anatomical landmarks, confirmed time of each lesion, ulcer, polyp visualised by the endoscopist, withdrawal time, mucosal inspection time, and complications (immediate and late: 24h post-procedure and 14 days post-procedure, respectively), the use of existing AI platforms that increase lesion detection (CADe) and classification (CADx), the AI classification (autonomous CADx diagnosis), the endoscopists' ODs without CADx, the endoscopists' ODs after seeing the diagnosis from CADx (CADx-assisted diagnosis), the performance of endoscopists (measured with detection rates such as ADR, AADR, SSLDR, PDR, or with detection counts such as APC). In the case of patients with rectal cancer, any active disease, such as tumor recurrence will be documented.

OTHER OUTCOMES:
Polyp, lesion, or ulcer-related characteristics | From enrollment to the end of histology assessment
  For upper and lower endoscopies, polyp, lesion, or ulcer-related characteristics will be documented: anatomical location, size estimated by the endoscopists, surface and vascular pattern and morphology. Any other pathological findings with the description of severity and anatomical location will be documented. Any biopsies taken during the procedure, and their location will be documented, including the number and a description of the biopsied tissue, as well as the reason for the biopsy.
IBD data | From enrollment to the end of the procedure
  In case of IBD indication, Crohn's disease and ulcerative colitis endoscopic characteristics will be graded and documented. The inflammation, ulceration/erosion, stricture, bleeding, and their related severity or extent in each colon segment will be documented. The endoscopic characteristics of the colon will also be documented, using components of the Mayo Score / DAI for Ulcerative Colitis, including vessels and bleeding.
Hiatal hernia data | From enrollment to the end of the procedure
  In case of hiatal hernia, the size of the hernia along with the related type will be documented.
GERD data | From enrollment to the end of the procedure
  In case of esophagitis (GERD), the Los Angeles classification of esophagitis will be used to define the grade and extent of the inflammation. The MUSE classification system will also be used to categorise esophageal lesions and strictures.
Barrett's esophagus data | From enrollment to the end the histology assessment
  In case of Barrett's esophagus, a detailed description of the esophagus will be documented: presence and extent of Barrett's esophagus, including the length of Barrett's segment in cm, the classification of Barrett's esophagus, the presence or absence of hiatal hernia and its size, and any sign of reflux esophagitis alongside their severity and location. The Prague classification will be used to describe the circumferential and maximal Barrett's segment length. The number and locations of biopsies taken within the Barrett's segment, at the GE junction, and in any suspicious area. The size and characteristics of any polyps or nodules found within the Barrett's segment will be documented as biopsies are essential for grading dysplasia and monitoring disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in research articles based on this video registry, after de-identification (text, tables, figures and appendices).
Access Criteria: Proposals should be directed to daniel.von.renteln.med@ssss.gouv.qc.ca . To gain access, data requestors will need to sign a data access agreement